CLINICAL TRIAL: NCT01650090
Title: Phase 2 Study of Inhaled Lipid Cisplatin in Pulmonary Recurrent Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eleison Pharmaceuticals LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EP-ILC-201
Record Dates: First submitted 2012-07-20; First posted 2012-07-26 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Relapse of Osteosarcoma
Keywords: Pulmonary relapse; Osteosarcoma; Lung metastases; Pediatric osteosarcoma; Inhaled chemotherapy; Inhaled Lipid Cisplatin
MeSH Terms: conditions — Osteosarcoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ILC (Experimental): Inhaled Lipid Cisplatin (ILC) will be administered every two weeks via nebulization and inhalation.
  Interventions: Drug: Inhaled Lipid Cisplatin (ILC)

INTERVENTIONS:
Drug: Inhaled Lipid Cisplatin (ILC) — ILC is provided as cisplatin in a lipid complex suspended in a saline solution. Every two weeks, the patient will receive 36 mg/m2 (measured as concentration of cisplatin) of ILC via nebulization. Treatment may continue for up to 1 year.
  Other Names: Cisplatin; Lipid cisplatin complex

SUMMARY:
To establish whether treatment with Inhaled Lipid Cisplatin (ILC) is effective in delaying/preventing pulmonary relapse in osteosarcoma patients in complete surgical remission following one or two prior pulmonary relapses.

DETAILED DESCRIPTION:
ILC is a novel formulation of cisplatin, designed for inhalation by nebulization. The anticipated pulmonary benefits of ILC over systemic cisplatin therapy are threefold:

* Increased local cisplatin concentrations
* Sustained release of cisplatin in the lungs
* Minimal systemic exposure to cisplatin

In this study, patients currently in surgical complete remission (CR) following one or two prior relapses of osteosarcoma involving pulmonary disease will be treated with ILC every two weeks for up to one year. ILC will be administered via nebulization.

ELIGIBILITY:
Inclusion Criteria:

1. History of osteosarcoma metastatic to the lung(s). (First or second pulmonary recurrence(s) removed by surgery, and previous second-line systemic chemotherapy is allowed).
2. Patients must be macroscopically disease free following pulmonary metastectomy of a single or multiple lesions. Complete remission surgically (free of macroscopic disease) is required. Pleural disruption and/or microscopic positive margins are allowed.
3. Age ≥13 years.
4. Patients must have recovered sufficiently from all acute adverse effects of prior therapies, excluding alopecia.
5. Patients must have an ECOG performance status of 0-2. (Lansky score of 50-100 if < 16 years old).
6. Patients must have recovered sufficiently from surgery and have adequate airflow and pulmonary reserve. This decision should be at the investigator's discretion taking into consideration pre-surgery pulmonary function. (As a guideline: adequate airflow defined by a measured Forced Expiratory Volume (FEV1) not less than 50% of the predicted value and adequate pulmonary reserve as evidenced by a FEV1/FVC ratio of 65% or greater).
7. Patients must have adequate renal function as defined by a serum creatinine of ≤ 1.5 mg/dl.
8. Patients must have adequate liver function as defined by total bilirubin of ≤ 1.5 mg/dl and ALT or AST < 2.5 times the institution's upper normal limit.
9. Patients must have adequate bone marrow function as defined by an absolute neutrophil count (ANC) of ≥ 1,000/mm3 and platelet count of ≥ 100,000/mm3.
10. Signed informed consent including, where applicable, the consent of the patient's legal guardian.

Exclusion Criteria:

1. Current extrapulmonary disease.
2. Current macroscopic pulmonary lesions.
3. Greater than 2 pulmonary recurrences.
4. Greater than 4 weeks since thoracotomy rendering patient free of macroscopic disease.
5. Females who are pregnant or breast-feeding.
6. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study.
7. Contraindication to or unwillingness to undergo multiple CT scans and chest X-rays.
8. Unwillingness or inability to comply with the study protocol for any other reason.
9. Participation in an investigational drug or device study or treatment with any anti-neoplastic agent within 14 days of the first day of dosing on this study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Observed Relapse Free Interval (RFI) | At relapse, estimated at 6-12 months average.
  Observed relapse free interval (RFI) will be compared to historical controls. Relapse free interval is defined as the time of diagnosis of the previous relapse to time of diagnosis of the new relapse.

SECONDARY OUTCOMES:
Median, 1, 2 and 5 year Overall Survival (OS) | 1, 2 and 5 Years
  The percentage of patients alive at 1, 2 and 5 years and the median overall survival.
Median, 1, 2 and 5 year Event Free Survival (EFS) | 1, 2 and 5 years
  The percentage of patients surviving without disease relapse at 1, 2 and 5 years and the median event free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gorlick, MD, Principal Investigator — The Children's Hospital at Montefiore; Forrest H Anthony, MD, PhD, Study Director — Eleison Pharmaceuticals
Locations (15):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington